CLINICAL TRIAL: NCT00620555
Title: A 52 Weeks, Open-Label, Multicenter Study Evaluating The Efficacy And Safety Of Gabapentin As Adjunctive Therapy In Pediatric Patients Who Have Completed The 12 Weeks Treatment In Study A9451162 (NCT00603473)
Brief Title: A Phase III Open-Label Extension Study Of Gabapentin As Adjunctive Therapy In Japanese Pediatric Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9451165
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2011-12-20 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2011-11

CONDITIONS: Epilepsies, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gabapentin (Experimental)
  Interventions: Drug: gabapentin

INTERVENTIONS:
Drug: gabapentin — Orally administered gabapentin

SUMMARY:
Examine the safety and efficacy of gabapentin as adjunctive therapy in Japanese pediatric patients with partial seizures

ELIGIBILITY:
Inclusion Criteria:

* Completion of study A9451162 (NCT00603473)

Exclusion Criteria:

* Seizures related to drugs or acute medical illness
* History of any serious medical or psychiatric disorder

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- Japan (22):
  - Pfizer Investigational Site, Obu-shi,Morioka-machi, Aichi-ken
  - Pfizer Investigational Site, Jonan-ku, Fukuoka
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Suma-Ku,Kobe, Hyōgo
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken
  - Pfizer Investigational Site, Zentsuuji, Kagawa-ken
  - Pfizer Investigational Site, Yokohama, Kanagawa Pref.
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Shōwaku, Nagoya
  - Pfizer Investigational Site, Niigata, Niigata
  - Pfizer Investigational Site, Kurashiki, Okayama Pref.
  - Pfizer Investigational Site, Okayama, Okayama-ken
  - Pfizer Investigational Site, Izumi-shi, Osaka
  - Pfizer Investigational Site, Miyakojima-ku, Osaka
  - Pfizer Investigational Site, Suita, Osaka
  - Pfizer Investigational Site, Shizuoka, Shizuoka
  - Pfizer Investigational Site, Kodaira, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Hiroshima
  - Pfizer Investigational Site, Saitama
  - Pfizer Investigational Site, Yamagata

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451165&StudyName=A%20Phase%20III%20Open-Label%20Extension%20Study%20Of%20Gabapentin%20As%20Adjunctive%20Therapy%20In%20Japanese%20Pediatric%20Patients%20With%20Partial%20Seizures

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Pediatric participants received gabapentin three times daily for 52 weeks. Participants aged 3 to 12 years received oral solution (250 mg/5 mL) at the dose calculated based on their body weight; 40 mg/kg/day for 3 to 4 years old and 25 to 35 mg/kg/day for 5 to 12 years old but not exceeding 1800 mg per day. Participants aged 13 to 15 years received gabapentin tablet at the dose of 1200 or 1800 mg/day. The dose was adjusted within the range of maintenance doses. Gabapentin could be increased if necessary with the maximum dose of 50 mg/kg/day for participants aged 3 to 12 years; All participants could receive gabapentin tablet not exceeding 2400 mg per day.
Period: Overall Study
Arm/Group | Gabapentin
Started | 65
Completed | 44
Not Completed | 21
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 2
Not completed — Lack of Efficacy | 12
Not completed — Withdrawal by Subject | 1
Not completed — Choice of other treatment | 1
Not completed — Visit failure against planned | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gabapentin
Number analyzed (Participants) | 65
Age, Customized [Number; unit: Participants]
  3-4 years | 8
  5-12 years | 42
  13-16 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities and Treatment-Related)
Description: Any untoward medical occurrence in a participant who received study drug was considered an adverse event (AE), without regard to possibility of causal relationship. Treatment-emergent adverse events: those which occurred or worsened after baseline. Severe AEs: those which interferes significantly with participant's usual function. An AE resulting in any of the following outcomes, was considered to be a serious adverse event: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect.
Time Frame: up to 53 weeks
Population: Safety analysis set: All paticipants who have received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Gabapentin
Number analyzed (Participants) | 65
Participants
  All-causality adverse events (AEs) | 58
  Treatment-related AEs | 13
  All-causality serious AEs | 2
  Treatment-related serious AEs | 0
  All-causality severe AEs | 1
  Treatment-related severe AEs | 0
  Discontinuation due to all-causality AEs | 4
  Discontinuation due to treatment-related AEs | 2
  Dose reduction due to all-causality AEs | 2
  Dose reduction due to treatment-related AEs | 2

2. Secondary Outcome: Response Ratio
Description: The Response Ratio calculated by the following equation : Response Ratio = (T minus B) divided by (T plus B), where T is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 52-week treatment period, and B is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 6-week baseline period of the previous study A9451162 (NCT00603473).
Time Frame: Up to 52 weeks
Population: Intent to treat (ITT): Subjects who have received at least one dose of the study drug and in whom the number of epileptic seizures used for efficacy assessment has been counted in both the baseline and treatment periods.
  n = number of participants who have total number of seizures at each assessment time point.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Gabapentin
Number analyzed (Participants) | 65
Ratio
  Week 1 to 8 (n=65) | -0.263 (0.3141)
  Week 9 to 16 (n=60) | -0.256 (0.3513)
  Week 17 to 24 (n=58) | -0.300 (0.3671)
  Week 25 to 36 (n=54) | -0.280 (0.3753)
  Week 37 to 52 (n=47) | -0.327 (0.3712)

3. Secondary Outcome: Responder Rate
Description: Responder Rate was defined as the percentage of subjects with a 50 percent or greater reduction in the seizure frequency per 28 days for the 52-week treatment period in comparison with the frequency per 28 days for the 6-week baseline period of the previous study A9451162 (NCT00603473).
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gabapentin
Number analyzed (Participants) | 65
Percentage of participants
  Week 1 to 8 (n=65) | 35.4 [23.9 to 48.2]
  Week 9 to 16 (n=60) | 40.0 [27.6 to 53.5]
  Week 17 to 24 (n=58) | 39.7 [27.1 to 53.4]
  Week 25 to 36 (n=54) | 40.7 [27.6 to 55.0]
  Week 37 to 52 (n=47) | 46.8 [32.1 to 61.9]

4. Secondary Outcome: Percent Change in Seizure Frequency
Description: Percent change in seizure frequency (PCH) was calculated as follows: PCH = 100*(T minus B) divided by B, where T is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 52-week treatment period, and B is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 6-week baseline period of the previous study A9451162 (NCT00603473).
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: Percent change
Arm/Group | Gabapentin
Number analyzed (Participants) | 65
Percent change
  Week 1 to 8 (n=65) | -34.2 [-100.0 to 63.1]
  Week 9 to 16 (n=60) | -33.0 [-100.0 to 99.8]
  Week 17 to 24 (n=58) | -42.0 [-100.0 to 112.5]
  Week 25 to 36 (n=54) | -41.6 [-100.0 to 110.7]
  Week 37 to 52 (n=47) | -49.2 [-100.0 to 131.7]

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Gabapentin
Serious Adverse Events (participants affected / at risk) | 2/65
Other Adverse Events (participants affected / at risk) | 48/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=65)
BRONCHOPNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1
ENCEPHALOPATHY (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=65)
Dental caries (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 8
Bronchitis (Infections and infestations) | 4
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 28
Pharyngitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Arthropod bite (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 4
Somnolence (Nervous system disorders) | 10
Eczema (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.